CLINICAL TRIAL: NCT05543564
Title: The Case for Selective Prophylactic Pan-retinal Photocoagulation in Moderate Non-Proliferative Diabetic Retinopathy in Ophthalmic Practice in Low- Resource Settings
Brief Title: Prophylactic PRP in Moderate NPDR
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdelazeem, Associate Professor, Assiut University
Other Study IDs: 17300819
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Eye Diseases; Diabetes; Diabetic Retinopathy
MeSH Terms: conditions — Eye Diseases; Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: PRP — Single session prophylactic early Pan-retinal Photocoagulation

SUMMARY:
Diabetic retinopathy (DR) is a challenge to ophthalmic practice in communities with poor socioeconomic development. The COVID 19 pandemic has accentuated the challenge. DR is one of the leading causes of vision loss worldwide, estimated to account for 1.25% of moderate to severe visual impairment and 1.07% of blindness. Pan retinal photocoagulation (PRP) remains the gold standard treatment for preventing visual loss in PDR. Scatter photocoagulation is not recommended for eyes with mild or moderate non-proliferative diabetic retinopathy (NPDR) provided careful follow-up can be maintained,. When retinopathy is more severe, scatter photocoagulation should be considered and should not be delayed if the eye has reached the high-risk proliferative stage. As many as 27% of patients with moderate NPDR are estimated to progress to PDR in 1 year; therefore, they should be seen every 4 to 8 months. This ideal, good as it is, is not what ophthalmic practice has to deal with in communities of low-resource settings, where patients often seek medical advice due to visual complaints from the complications of PDR without being diagnosed in the non-proliferative stage or high risk PDR. Screening protocols are not followed, a situation aggravated during the COVID pandemic lockdown.

ELIGIBILITY:
Inclusion Criteria:

Patients with moderate NPDR at high risk which includ:

* Patients with PDR in the other eye
* Patients whose Glycosylated Haemoglobin (HbA1c) more than 8 %.
* Patients with early cataract
* Patients on regular renal dialysis or with impaired renal function
* Patients with restricted mobility because of neurological or orthopedic conditions
* Patients dependent on others, including old age.
* Women in rural areas, who are dependent on the accompaniment of a male relative.

Exclusion Criteria:

* Any patient who or whose relatives confirmed their attendance for regular follow-up according to the planned schedules after being informed of the possible complications which could happen if he or she did not attend.
* Patients with clinically significant macular edema (CSME).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate NPDR at high risk
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
BCVA | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt